CLINICAL TRIAL: NCT04213898
Title: SHR-1210 Combined With Albumin-bound Paclitaxel and Epirubicin Neoadjuvant for Triple Negative Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wachengzheng, Doctor, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-TNBC-HN100
Record Dates: First submitted 2019-12-27; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Epirubicin; camrelizumab; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210+Albumin-bound paclitaxel+Epirubicin (Experimental): Neoadjuvant therapy：SHR-1210+Albumin-bound paclitaxel+Epirubicin
  Interventions: Drug: SHR-1210+Albumin-bound paclitaxel + epirubicin

INTERVENTIONS:
Drug: SHR-1210+Albumin-bound paclitaxel + epirubicin — Neoadjuvant therapy：SHR-1210, 200mg,iv, q3w, for 6 cycles; Albumin-bound paclitaxel: 125 mg/m2, iv, d1, d8, and d15, 21 days as a cycle, for 6 cycles; Epirubicin: 75mg / m2, iv, d1, 21 days as a cycle, for 6 cycles; The surgery was performed 3-4 weeks after the completion of neoadjuvant chemotherapy.
  Other Names: camrelizumab for injection

SUMMARY:
Triple negative breast cancer (TNBC), characterized by estrogen receptor, progesterone receptor and HER2 negative, accounts for 10-20% of all breast cancers and usually occurs in young women. It is an aggressive and worst prognosis breast cancer subtype, which urgently requires effective treatment.The pathological complete response (pCR) of neoadjuvant therapy is associated with disease-free survival (DFS) and overall survival (OS) of breast cancer. The correlation between pathological response and long-term survival in patients with early-stage breast cancer is the strongest among patients with triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Newly treated female patients aged ≥18 years and ≤60 years; 2. ECOG score 0 ~ 1 points; 3. Pathologically confirmed, the core biopsy of breast tumor lesions identified patients with TNBC breast cancer; Note: ER and PR negatives are defined as ≤ 10% of cells expressing hormone receptors by IHC (immunohistochemistry) analysis. HER2 (human epidermal growth factor receptor 2) negative is defined as any of the following assessments: non-amplified in situ hybridization (ISH) (ratio ≤ 2.2), or IHC 0 or IHC 1+; 4. Evaluate measurable tumor lesions by ultrasound or magnetic resonance imaging (MRI) within 21 days before enrollment, size ≥2cm; 5. The main organs function normally, that is, they meet the following criteria:

  1. Blood routine examination standards must meet: ANC ≥1.5 × 109 / L; PLT ≥90 × 109 / L; Hb ≥90g / L;
  2. Biochemical examination must meet the following standards: TBIL ≤ upper limit of normal value (ULN); ALT and AST ≤ 1.5 times the upper limit of normal value (ULN); alkaline phosphatase ≤ 2.5 times the upper limit of normal value (ULN); BUN and Cr ≤ 1.5 × ULN and creatinine clearance ≥50 mL / min (CockcroftGault formula);
  3. The coagulation test standard must meet: the international standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN, and the activated partial thromboplastin time (aPTT) ≤ 1.5x ULN;
  4. Color Doppler ultrasound and echocardiography: left ventricular ejection fraction (LVEF≥55%);
  5. 18-lead electrocardiogram Fridericia-corrected QT interval (QTcF) for women <470 ms; 6. No evidence of distant metastases, including bilateral mammograms, breast ultrasounds; 7. Provide core biopsies from tumor lesions before treatment begins to confirm TNBC status and biomarker analysis; 8. For women who are not menopausal or not undergoing surgical sterilization: agree to abstinence or use an effective method of contraception during treatment and at least 7 months after the last dose during study treatment; 9. Sign the informed consent.

Exclusion Criteria:

* 1. Inflammatory breast cancer or stage IV (metastatic) breast cancer; 2. Have previously been treated with anti-PD-1, anti-PD-L1, anti-PD-L2 drugs or drugs that target another co-inhibitory T cell receptor (eg CTLA-4, OX-40, CD137); 3． Have previously received antitumor treatment or radiation therapy for any malignant tumor, excluding cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma; 4． Also receiving anti-tumor therapy in other clinical trials, including endocrine therapy, bisphosphate therapy or immunotherapy; 5. Have undergone major breast cancer-free surgery within 4 weeks before enrollment, or the patient has not fully recovered from such surgery; 6. Severe heart disease or discomfort, including but not limited to the following:

  --A history of diagnosis of heart failure or systolic dysfunction (LVEF <50%)
* High-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate> 100 bpm, significant ventricular arrhythmias (such as ventricular tachycardia) or higher-level atrioventricular block (ie Mobitz II second-degree atrioventricular block or third-degree atrioventricular block)

  --Angina pectoris requiring antianginal medication
* Clinically significant heart valve disease

  --ECG shows transmural myocardial infarction
* Poorly controlled hypertension (systolic blood pressure> 180 mmHg and / or diastolic blood pressure> 100 mmHg); 7. Have an autoimmune disease or other disease that requires systemic treatment with corticosteroids or immunosuppressive drugs (physical corticosteroid replacement therapy that allows adrenal or pituitary insufficiency); 8. A history of primary or acquired immunodeficiency (including allograft transplantation); 9. Female patients during pregnancy and lactation, female patients with fertility and a positive baseline pregnancy test, or women of childbearing age who are unwilling to take effective contraception during the entire trial and within 7 months after the last study medication; 10. have a history of (non-infectious) pneumonia, or currently have pneumonia that requires steroid therapy; 11. Active or previously documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis); 12. Known medical history of the following infections:

  * Human Immunodeficiency Virus (HIV)
  * A history of acute or chronic hepatitis B or C
* Received live virus vaccine within 30 days of planned start of treatment. Allow use of seasonal influenza vaccines that do not contain live viruses; 13. People with a known history of allergies to the drug components of this program; a history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; 14. Suffering from a serious concomitant disease or other comorbid condition that interferes with the planned treatment, or any other condition that the investigator considers the patient unsuitable to participate in this study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | At time of surgery
  TpCR (ypT0 / is, ypN0) assessed by pathologists participating in the research center: defined as the pathological evaluation of hematoxylin and eosin-stained resected breast cancer samples and all ipsilateral lymph node samples after neoadjuvant therapy and surgery there is any residual invasive cancer.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | up to 2 year
  Time after R0 resection to disease recurrence or death Time after R0 resection to disease recurrence or death Time after R0 resection to disease recurrence or death Defined as the time interval from the first day of disease-free (ie, the date of surgery) to the first recording of related events, which include recurrence of postoperative disease and death from any cause
Objective Response Rate (ORR) | up to 1 year
  CR+PR